CLINICAL TRIAL: NCT04982003
Title: Feasibility and Effects of Whole-body Drumming Classes on Walking in People With Parkinson's Disease: a Pilot Study
Brief Title: Feasibility of Whole-body Drumming Classes for People With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.T. Still University of Health Sciences (Other)
Responsible Party: Principal Investigator, Tara McIsaac, Principal Investigator, A.T. Still University of Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-004
Record Dates: First submitted 2021-05-18; First posted 2021-07-29 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: single group, pre- post-test design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group (Experimental): A single group of subjects with pretest, posttest, and one-month follow-up testing relative to 10-week drumming exercise classes
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — 10 weekly hour-long classes of drumming to music using large-amplitude, whole-body movements

SUMMARY:
People with Parkinson's disease (PD) experience difficulty with gait, postural instability, and lack of movement coordination and rhythmic timing. Non-motor functions affected by PD include time perception, feelings of apathy, depression, decreased self-efficacy, and decrease self-reported quality of life. There is currently a lack of information on how a therapeutic drumming class that uses whole-body large-amplitude movements to music would impact these motor and non-motor impairments in individuals with PD. The primary purpose of this study is to assess the feasibility of a 10-week whole-body drumming class to music specifically selected for its rhythmic structure, and effects on movement rhythm and time perception in individuals with PD. The secondary purpose is to assess the effects of the drumming class on apathy, depression, self-efficacy and health-related quality of life. Participants will be included if they have a diagnosis of PD and are able to move for an hour with rests, either standing or seated. Participants are tested before and after the class series and one month following.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with PD
* independent walking short community and household distances with or without assistive device
* able to participate in a 1-hour class once a week for ten weeks

Exclusion Criteria:

* change of Parkinson's medication or deep brain stimulation parameters within 2 weeks prior to or during the study
* inability to grasp 2-inch diameter "drum sticks"
* any conditions with contraindications to lift upper extremities overhead
* any medical restrictions to exercise

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Step Cadence Variability | within 7 days before the intervention
  Variability (SD) of step cadence
Step Cadence Variability | within 7 days after intervention
  Variability (SD) of step cadence
Step Cadence Variability | 1-month following intervention
  Variability (SD) of step cadence
Stride Length Variability | within 7 days before the intervention
  Variability (SD) of stride length
Stride Length Variability | within 7 days after intervention
  Variability (SD) of stride length
Stride Length Variability | 1-month following intervention
  Variability (SD) of stride length
Change in repeated finger-tapping | within 7 days before the intervention and within 7 days after intervention
  change in inter-tapping intervals (ms) change from pre- to post-intervention
Change in repeated finger-tapping | within 7 days before the intervention and 1-month following end of intervention
  change in inter-tapping intervals (ms) change from pre- to 1-month following end of intervention

SECONDARY OUTCOMES:
Change in Nine-hole peg test (NHP) duration (s) | within 7 days before the intervention and within 7 days after intervention
  change in speed of manual dexterity (s on NHP) from pre- to post-intervention
Change in Nine-hole peg test (NHP) duration (s) | within 7 days before the intervention, and 1-month following intervention
  change in speed of manual dexterity (s on NHP) from pre- to 1-month following end of intervention
Change in Physical Performance Test (PPT) score | within 7 days before the intervention and within 7 days after intervention
  change in whole-body functional mobility (PPT score; 0-36; higher is better) from pre- to post-intervention.
Change in Physical Performance Test (PPT) score | within 7 days before the intervention, and 1-month following intervention
  change in whole-body functional mobility (PPT score; 0-36; higher is better) from pre- to 1-month following end of intervention
Change in Parkinson Disease Questionnaire (PDQ-39) | within 7 days before the intervention and within 7 days after intervention
  change in disease-related quality of life (PDQ-39 score; 0-100, lower is better with improved quality of life) from pre- to post-intervention
Change in Parkinson Disease Questionnaire (PDQ-39) | within 7 days before the intervention, and 1-month following intervention
  change in disease-related quality of life (PDQ-39 score; 0-100, lower is better with improved quality of life) from pre- to 1-month following end of intervention
Geriatric Depression Scale (GDS) | within 7 days before the intervention and within 7 days after intervention
  change in depression (GDS score; 0-15, higher is worse with more depression) from pre- to post-intervention
Geriatric Depression Scale (GDS) | within 7 days before the intervention, and 1-month following intervention
  change in depression (GDS score; 0-15, higher is worse with more depression) from pre- to 1-month following end of intervention
General Self-Efficacy scale (GSE) | within 7 days before the intervention and within 7 days after intervention
  change in self-efficacy (GSE score; 10-40, higher is better with more self-efficacy) from pre- to post-intervention
General Self-Efficacy scale (GSE) | within 7 days before the intervention, and 1-month following intervention
  change in self-efficacy (GSE score; 10-40, higher is better with more self-efficacy) from pre- to 1-month following end of intervention
Lille Apathy Rating Scale (LARS) | within 7 days before the intervention and within 7 days after intervention
  change in apathy (LARS score; -36 to +36, lower is better with less apathy) from pre- to post-intervention
Lille Apathy Rating Scale (LARS) | within 7 days before the intervention, and 1-month following intervention
  change in apathy (LARS score; -36 to +36, lower is better with less apathy) from pre- to 1-month following end of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Tara L McIsaac, PhD, PT, Principal Investigator — A.T. Still University
Locations (1):
- A.T. Still University Arizona School of Health Sciences, Mesa, Arizona, United States

IPD SHARING:
Plan to Share IPD: No